CLINICAL TRIAL: NCT00000340
Title: Pemoline in the Treatment of Stimulant Dependence
Brief Title: Pemoline in the Treatment of Stimulant Dependence - 5
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never funded.
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-3-0010-5; Y01-3-0010-5
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Pemoline

INTERVENTIONS:
Drug: Pemoline

SUMMARY:
The purpose of this study is to assess the efficacy of pemoline in treating cocaine and/or methamphetamine dependent adults with comorbid Adult Attention Deficit Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Meet DSM-IV criteria for cocaine dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nuring women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical condtions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 1996-06

PRIMARY OUTCOMES:
Retention
Depression
Incidence of stimulant use
Severity of stimulant withdrawal symptoms
ADHD symptom severity
Degree of drug craving
Frequency of IV drug use and sexual risk behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.